CLINICAL TRIAL: NCT03660189
Title: The "Two Bag" System for Treatment of Adults With Diabetic Ketoacidosis: a Prospective Randomized Study
Brief Title: Two Bag System for Diabetic Ketoacidosis
Acronym: 2BagDKA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID19 restrictions impeded our ability to recruit patients further
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Vidya Krishnan, Professor, Case Western Reserve University, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB18-00025
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Ketoacidosis
Keywords: intravenous fluids; adults; two bag system
MeSH Terms: conditions — Diabetic Ketoacidosis | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Usual care with a one bag system of IV fluids, as recommended in the American Diabetes Association consensus statement guidelines from 2009.
- Two bag system (Experimental): A two bag system of IV fluids will be used during insulin infusion administration.
  Interventions: Other: Two bag system

INTERVENTIONS:
Other: Two bag system — The two IV fluid bags have identical fluids and electrolytes, except one has 10% dextrose and the other has no dextrose. The two fluid bags run simultaneously and their rates are adjusted according to the patient's blood sugar.
  Arms: Two bag system

SUMMARY:
This is a study investigating the best way to treat diabetic ketoacidosis (DKA) with intravenous (IV) fluids in the hospital. The purpose of this study is to determine whether the "two bag" system of administering IV fluids for the treatment of adults with DKA leads to a shorter time requiring intravenous insulin (a shorter time to anion gap closure), when compared to usual care the traditional "one bag" system of IV fluids. Participants will be assigned randomly to either the usual care group or the "two bag" system group. Based on studies performed in the past, the investigators predict that patients treated with the two bag system of IV fluids for DKA will have a significantly shorter time requiring treatment with intravenous insulin when compared to the traditional one bag system.

DETAILED DESCRIPTION:
The two bag system has been studied in the pediatric population and is used frequently in pediatric intensive care units. It involves two bags of identical fluids with electrolytes, except one bag has 0% dextrose and the other has 10% dextrose. The two fluid bags run simultaneously into a single IV. The rates of the two fluid bags are adjusted according to the patient's blood sugar. Since the hyperglycemia in DKA typically corrects before the ketosis, this provides a more efficient method of titrating the dextrose concentration based on the patient's needs, while continuing to infuse the insulin at a constant rate to prevent further ketogenesis. The benefits of the two bag system from the pediatric literature include: decreased response time to IV fluid changes, decreased time to correction of bicarbonate and ketones, and decreased total IV fluid volume administered. There was one retrospective study of the two bag system in adults, which showed decreased time to anion gap closure and decreased hypoglycemic events. To this date, there are no prospective randomized trials to evaluate the efficacy of the two bag system in adults.

Patients admitted with DKA in the critical care pavilion will be randomized to either the "two bag system" or "usual care" group.

Patients in both groups will be treated for DKA with IV fluid resuscitation for dehydration and an insulin infusion according to usual care, recommended at 0.1 U/kg/hr.

The two bag system of IV fluids will be ordered as delineated below:

If blood sugar is > 300, run D10 solution at 0 ml/hr and saline solution at 200 ml/hr.

If blood sugar is 250-299, run D10 solution at 50 ml/hr and saline solution at 150 ml/hr.

If blood sugar is 200-249, run D10 solution at 100 ml/hr and saline solution at 100 ml/hr.

If blood sugar is 150-199, run D10 solution at 150 ml/hr and saline solution at 50 ml/hr.

If blood sugar is < 150, run D10 solution at 200 ml/hr and saline solution at 0 ml/hr.

The control group will be usual care of DKA based on the American Diabetes Association Guidelines using a "one bag system."

In both groups, blood sugars will be checked every hour while on the insulin drip. A basic metabolic panel will be checked every 4 hours to monitor the anion gap. Once the anion gap is closed on two occasions and the subject is able to tolerate an enteral diet, the patient will be transitioned to subcutaneous insulin and insulin drip will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of diabetic ketoacidosis defined as:

   1. Blood sugar greater than 250 mg/dl
   2. Venous pH less than 7.25
   3. Bicarbonate less than 18
   4. Evidence of ketone formation with either positive urine ketones or elevated beta-hydroxybutyrate > 3
   5. Anion gap greater than 10 +/ - 2 (or higher than expected anion gap corrected for albumin)
2. 18-85 years of age

Exclusion Criteria:

1. Pregnancy
2. Hyperglycemic hyperosmolar state
3. Ketosis from other etiology such as starvation or alcoholic ketosis
4. Acute exacerbation of congestive heart failure
5. Acute coronary syndrome or non-ST elevation MI
6. Pulmonary edema from other cause such as decompensated liver failure or acute renal failure
7. Renal failure requiring renal replacement therapy (hemodialysis)
8. Septic shock

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vidya Krishnan, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share individual participant data at this time.

REFERENCES:
- [Background] Kitabchi AE, Umpierrez GE, Murphy MB, Kreisberg RA. Hyperglycemic crises in adult patients with diabetes: a consensus statement from the American Diabetes Association. Diabetes Care. 2006 Dec;29(12):2739-48. doi: 10.2337/dc06-9916. No abstract available. PMID 17130218
- [Background] Grimberg A, Cerri RW, Satin-Smith M, Cohen P. The "two bag system" for variable intravenous dextrose and fluid administration: benefits in diabetic ketoacidosis management. J Pediatr. 1999 Mar;134(3):376-8. doi: 10.1016/s0022-3476(99)70469-5. PMID 10064682
- [Background] So TY, Grunewalder E. Evaluation of the two-bag system for fluid management in pediatric patients with diabetic ketoacidosis. J Pediatr Pharmacol Ther. 2009 Apr;14(2):100-5. doi: 10.5863/1551-6776-14.2.100. PMID 23055897
- [Background] Munir I, Fargo R, Garrison R, Yang A, Cheng A, Kang I, Motabar A, Xu K, Loo LK, Kim DI. Comparison of a 'two-bag system' versus conventional treatment protocol ('one-bag system') in the management of diabetic ketoacidosis. BMJ Open Diabetes Res Care. 2017 Aug 11;5(1):e000395. doi: 10.1136/bmjdrc-2017-000395. eCollection 2017. PMID 28878933
- [Background] Poirier MP, Greer D, Satin-Smith M. A prospective study of the "two-bag system'' in diabetic ketoacidosis management. Clin Pediatr (Phila). 2004 Nov-Dec;43(9):809-13. doi: 10.1177/000992280404300904. PMID 15583776

RESULTS

PARTICIPANT FLOW:
Groups:
- Two Bag System: A two bag system of IV fluids will be used during insulin infusion administration.
  Two bag system: The two IV fluid bags have identical fluids (normal saline or half normal saline) and electrolytes (optional addition of potassium chloride or potassium phosphate), except one has 10% dextrose and the other has no dextrose. The two fluid bags run simultaneously and their rates are adjusted according to the patient's blood sugar. Total fluid rate (sum of rates of two bags) is 200mL/hour.
Period: Overall Study
Arm/Group | Usual Care | Two Bag System
Started | 25 | 32
Completed | 25 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Two Bag System | Total
Number analyzed (Participants) | 25 | 32 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (13.3) | 38.6 (13.6) | 37.1 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 21 | 36
  Male | 10 | 11 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 32 | 57
Type of Diabetes (Number of Participants with Type 1 DM) [Count of Participants; unit: Participants] | 20 | 19 | 39
pH on VBG (venous blood gas) at time of presentation [Mean (Standard Deviation); unit: unitless] — range from 0 to 14, 7.0 is neutral Population: Initial VBG unavailable for 1 participant in the usual care group.
  unitless
    number analyzed (Participants) | 24 | 32 | 56
    (all) | 7.11 (0.14) | 7.09 (0.14) | 7.10 (0.14)

OUTCOME MEASURES:

1. Primary Outcome: Time to Anion Gap Closure in Hours
Description: Anion gap (Na - Cl - HCO3) is within normal range when corrected for the albumin (time to anion gap closure will be defined as the time to the first occurrence of a normal anion gap).
Time Frame: while in DKA
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Usual Care | Two Bag System
Number analyzed (Participants) | 25 | 32
hours
  Time to AG closure (from ED admit) | 11.2 (5.1) | 12.2 (3.9)
  Time to AG closure (from first BMP) | 12.0 (6.7) | 13.5 (7.7)
Statistical Analysis 1: Comparison: Usual Care vs Two Bag System; Test type: Superiority; p = 0.54, t-test, 2 sided
Statistical Analysis 2: Comparison: Usual Care vs Two Bag System; Test type: Superiority; p = 0.44, t-test, 2 sided

2. Secondary Outcome: Number of Participants Experiencing Hypoglycemic Episodes
Description: Symptomatic episodes of hypoglycemia
Time Frame: while in DKA
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Two Bag System
Number analyzed (Participants) | 25 | 32
Participants | 0 | 0

3. Secondary Outcome: Number of Participants Experiencing Hypoxic Episodes
Description: Desaturations less than 89% requiring supplemental oxygen
Time Frame: while in DKA
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Two Bag System
Number analyzed (Participants) | 25 | 32
Participants | 0 | 1
Statistical Analysis 1: Comparison: Usual Care vs Two Bag System; Test type: Superiority; p = 1.0, Fisher Exact

4. Secondary Outcome: Pulmonary Edema
Description: Pulmonary edema seen on either chest X-ray or with the change in the lung exam
Time Frame: while in DKA
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Two Bag System
Number analyzed (Participants) | 25 | 32
Participants | 0 | 0

5. Secondary Outcome: Chest Pain With EKG Changes
Description: Onset of new chest pain with new EKG changes concerning for ischemia
Time Frame: while in DKA
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Two Bag System
Number analyzed (Participants) | 25 | 32
Participants | 0 | 0

6. Secondary Outcome: Hyponatremia Events
Description: Sodium values less than 135 mmol/L (corrected for glucose)
Time Frame: while in DKA
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Two Bag System
Number analyzed (Participants) | 25 | 32
Participants | 9 | 12
Statistical Analysis 1: Comparison: Usual Care vs Two Bag System; Test type: Superiority; p = 0.91, Fisher Exact

7. Secondary Outcome: Hypokalemia Events
Description: Potassium values less than 3.3 mmol/L
Time Frame: while in DKA
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Two Bag System
Number analyzed (Participants) | 25 | 32
Participants | 2 | 5
Statistical Analysis 1: Comparison: Usual Care vs Two Bag System; Test type: Superiority; p = 0.45, Fisher Exact

8. Secondary Outcome: ICU Length of Stay
Description: Total time the patient was admitted in the stepdown unit and/or medical ICU
Time Frame: during hospitalization
Reporting Status: Not Posted

9. Secondary Outcome: Changes in Mental Status
Description: Worsening in either CAM-ICU score or Glasgow Coma Scale
Time Frame: while in DKA
Reporting Status: Not Posted

10. Secondary Outcome: Total Volume of Intravenous Fluids Administered
Description: Total volume of intravenous fluids administered
Time Frame: while in DKA
Reporting Status: Not Posted

11. Secondary Outcome: Hypernatremia
Description: Maximum sodium level > 153 mmol/L
Time Frame: while in DKA
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Two Bag System
Number analyzed (Participants) | 25 | 32
Participants | 1 | 2
Statistical Analysis 1: Comparison: Usual Care vs Two Bag System; Test type: Superiority; p = 1.0, Fisher Exact

12. Secondary Outcome: Hyperkalemia
Description: Maximum K level > 5.3 mmol/L
Time Frame: while in DKA
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Two Bag System
Number analyzed (Participants) | 25 | 32
Participants | 3 | 5
Statistical Analysis 1: Comparison: Usual Care vs Two Bag System; Test type: Superiority; p = 1.0, Fisher Exact

ADVERSE EVENTS:
Time Frame: During the index hospitalization - from time of onset of DKA (time of ED check-in or time of first BMP, whichever is first) through the resolution of the DKA. This would be an average of about 12 hours, and a maximum of 48.5 hours.
Description: Review of EMR
Arm/Group | Usual Care | Two Bag System
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/32
Other Adverse Events (participants affected / at risk) | 0/25 | 0/32

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed (due to COVID19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT03660189/Prot_SAP_000.pdf